CLINICAL TRIAL: NCT00002050
Title: A Study of Thymopentin Effects on HIV-1 Infectivity of Blood Mononuclear Cells and Semen in HIV Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Immunobiology Research Institute (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 015D; H87-75
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-08

CONDITIONS: HIV Infections
Keywords: Semen; Thymopentin; Leukocytes, Mononuclear; AIDS-Related Complex
MeSH Terms: conditions — HIV Infections; AIDS-Related Complex | interventions — Thymopentin

INTERVENTIONS:
Drug: Thymopentin

SUMMARY:
Examine the ability of Timunox (thymopentin) to reduce the amount and/or frequency of virus isolation. Examine the ability of thymopentin to stimulate the immune system and alter the clinical findings in patients infected with HIV who do not yet have AIDS.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Aerosolized pentamidine.

Patients must have the following:

* Seropositive for HIV-1 (ELISA assay) confirmed by Western blot.
* HIV-1 p24 antigen must be detected in supernatant fluids from co-cultures of patients' PBMC on two separate occasions.
* Voluntarily sign consent.
* Patients with HIV "wasting syndrome" are allowed.

Prior Medication:

Allowed:

* Aerosolized pentamidine.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* AIDS as defined by the CDC.
* Significant hepatic disease.
* Thrombocytopenia.
* Hypersensitivity to thymopentin.
* Hemophilia A or B or other hematologic disorders requiring current or previous administration of blood products.
* Abnormal chest x-ray (indicative of active disease (opportunistic infection)) within 30 days prior to study entry.

Patients with the following are excluded:

* AIDS as defined by the CDC.
* Significant hepatic disease.
* Thrombocytopenia.
* Hypersensitivity to thymopentin.
* Hemophilia A or B or other hematologic disorders requiring current or previous administration of blood products.
* Abnormal chest x-ray (indicative of active disease (opportunistic infection)) within 30 days prior to study entry.

Prior Medication:

Excluded within 30 days of study entry:

* Immunomodulatory or experimental therapy.
* Excluded within 90 days of study entry:
* Zidovudine (AZT).

Intravenous drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Immunobiology Research Institute, Annandale, New Jersey, United States